CLINICAL TRIAL: NCT03851549
Title: US Regulatory Clinical Evaluation - User Performance and System Use Evaluation of a New Blood Glucose Monitoring System.
Brief Title: A User Performance and System Use Evaluation of a New Blood Glucose Monitoring System ( BGMS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LifeScan Scotland Ltd (Industry)
Collaborators: Institut für Diabetes-Technologie ( IfDT) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3178226
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Blood Glucose monitoring System (BGMS) (Experimental): Intervention: Blood Glucose monitoring Systems (BGMS): Results obtained from the new BGMS for UP are compared to a reference instrument (YSI 2300)
  Interventions: Device: New BGMS (US)

INTERVENTIONS:
Device: New BGMS (US) — New blood glucose monitoring system / In vitro diagnostic device (IVDD)

SUMMARY:
This study is the US Regulatory Clinical Evaluation - User Performance and System Use Evaluation of a new Blood Glucose Monitoring System (BGMS).

DETAILED DESCRIPTION:
User Performance - Assess Lay User fingertip test results obtained on the new BGMS compared to a validated method (YSI 2300 STAT PLUS glucose analyzer results) according to FDA Guidance 2016 section VI.C.

Assess System Use of the new BGMS, as relevant to self-testing technique, with reference to the Owner's Booklet.

ELIGIBILITY:
Summary of inclusion criteria:

Subject is at least 12 years old. Informed Consent. Subject has a current diagnosis of type 1 or type 2 diabetes mellitus. Subject reads and understands English. Subject is currently performing unassisted self-monitoring of blood glucose (SMBG) OR naive to SMBG for a 10% sub-group.

Summary of exclusion criteria:

Conflict of interest. Technical expertise.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2019-03-12 (Estimated); Primary Completion 2019-04-19 (Estimated); Study Completion 2019-04-19 (Estimated)

PRIMARY OUTCOMES:
User Performance ( UP) | < 30 minutes
  User Performance evaluation (referred to as Method Comparison / User Evaluation in FDA Guidance 2016): Lay User accuracy of BGMS by comparison of meter blood glucose results to a laboratory reference instrument.
System Use Evaluation | < 30 minutes
  System usability: Lay user system use evaluation (as relevant to fingertip self-testing) by study personnel observation and completion of a scoring questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Macleod, Study Director — LifeScan Scotland
Locations (4):
- Institut für Diabetes-Technologie, Ulm, Germany
- United Kingdom (3):
  - Royal Infirmary of Edinburgh, Edinburgh, Lothian
  - Birmingham Heartlands Hospital, Birmingham
  - Centre for Health Science, Inverness

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Katz LB, Stewart L, King D, Cameron H. Meeting the New FDA Standard for Accuracy of Self-Monitoring Blood Glucose Test Systems Intended for Home Use by Lay Users. J Diabetes Sci Technol. 2020 Sep;14(5):912-916. doi: 10.1177/1932296820906184. Epub 2020 Feb 14. PMID 32059615